CLINICAL TRIAL: NCT06874816
Title: Does Your Jaw Tell the Story of Your Pain? Masseter Muscle Thickness, Bruxism, and Oral Behaviors in Chronic Non-Specific Neck Pain
Brief Title: Masseter Thickness, Bruxism, and Oral Behaviors in Chronic Neck Pain
Status: Recruiting | Type: Observational
Sponsor: Beylikduzu State Hospital (Other)
Responsible Party: Principal Investigator, Busra Sirin, MD, Beylikduzu State Hospital
Other Study IDs: Beylikdüzüstateh14
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Neck Pain
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neck pain group: Patients with chronic non specific neck pain
- Healthy controls: Healthy controls

SUMMARY:
A total of 30 patients aged 18-65 years who present with chronic non-specific neck pain and 30 healthy volunteers will be included in the study. Patients with symptoms persisting for at least 3 months will be eligible for inclusion. Necessary information will be provided to all participants, and informed consent will be obtained.

To assess pain severity before treatment, participants will be asked to rate their complaints using the Visual Analog Scale (VAS), a linear scale for pain assessment. The Neck Disability Index will be used to determine the level of disability.

The Jaw Functional Limitation Scale-20 (JFLS-20), Patient Health Questionnaire-9 (PHQ-9), Patient Health Questionnaire-15: Physical Symptoms, Generalized Anxiety Disorder-7 (GAD-7), and the Oral Behaviors Checklist-included in Axis 2 of the DC/TMD form developed for evaluating temporomandibular joint dysfunction-will be used to assess patients' psychosocial characteristics and parafunctional habits.

Additionally, masseter muscle thickness will be evaluated using ultrasonographic measurement.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with chronic non-specific neck pain
* Aged between 18-65 years
* Symptoms persisting for at least 3 months

Exclusion Criteria:

* Pregnancy
* Presence of psychiatric or neurological diseases
* Use of psychiatric medications
* Cognitive impairment
* History of neck injection or surgery within the last 6 months
* Presence of rheumatic diseases
* Spinal stenosis
* Cervical disc herniation
* Advanced degeneration detected in radiological imaging
* History of fracture or surgery in the temporomandibular joint
* Presence of inflammatory, rheumatologic diseases, or malignancy affecting the t--emporomandibular joint

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study population will consist of 30 patients diagnosed with chronic non-specific neck pain and 30 healthy volunteers, aged between 18 and 65 years.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2025-03-10 (Actual); Primary Completion 2025-04-10 (Estimated); Study Completion 2025-04-10 (Estimated)

PRIMARY OUTCOMES:
Masseter Muscle Thickness | 0 day
  Measured using ultrasonography, with values interpreted in relation to clinical findings. No fixed score range; thickness is recorded in millimeters.

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) | 0 day
  A linear scale used to assess pain severity, where higher scores indicate more severe pain. Score range: 0-10.
Neck Disability Index | 0 day
  A questionnaire used to evaluate the level of disability related to neck pain, with higher scores reflecting greater disability. Score range: 0-100.
Patient Health Questionnaire-9 (PHQ-9) | 0 day
  A scale measuring the severity of physical symptoms, where higher scores represent greater somatic symptom burden. Score range: 0-30.
Generalized Anxiety Disorder-7 (GAD-7) | 0 day
  A scale used to assess anxiety levels, with higher scores indicating more severe anxiety symptoms. Score range: 0-21.
Jaw Functional Limitation Scale-20 (JFLS-20) | 0 day
  A tool used to evaluate functional limitations of the jaw, where higher scores indicate greater impairment. Score range: 0-100.
Oral Behaviors Checklist | 0 day
  A questionnaire used to identify parafunctional oral habits, with higher scores reflecting more frequent parafunctional activities. No predefined score range; higher scores indicate greater frequency.

CONTACTS AND LOCATIONS:
Locations (1):
- Beylikdüzü State Hospital, Istanbul, Beylikdüzü, Turkey (Türkiye)